CLINICAL TRIAL: NCT03450057
Title: Efficacy of Daratumumab in Patients With Relapsed/Refractory Myeloma With Renal Impairment
Acronym: DARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAE-2017/MM02; 2017-003950-18 (EudraCT Number)
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2022-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Multiple Myeloma; MM; Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab; Dexamethasone; darlin protein, Dictyostelium

STUDY DESIGN:
Intervention Model Description: Single arm: Daratumumab and Dexamethasone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm trial receiving daratumumab with dexamethasone (DaraD) (Experimental): Daratumumab was given at a dose of 16 mg/kg administered as an intravenous (IV) infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Dexamethasone was administered according to the standard recommended dose of 40 mg (20 mg for patients > 75 years of age) orally once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
  Interventions: Drug: Daratumumab with dexamethasone

INTERVENTIONS:
Drug: Daratumumab with dexamethasone — Daratumumab:
  Daratumumab was given at a dose of 16 mg/kg administered as an intravenous (IV) infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects received pre-infusion medications before infusions to mitigate potential infused-related reactions (IRRs).
  Dexamethasone:
  Dexamethasone was administered at 40 mg (20 mg for patients >75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
  Other Names: DaraD; Darzalex; Dara; Dex

SUMMARY:
The purpose of this study was to evaluate the effects of daratumumab with dexamethasone (DaraD) in subjects with relapsed or refractory multiple myeloma and renal impairment.

DETAILED DESCRIPTION:
This was a multicenter, single arm, open-label phase 2 study. 38 subjects were enrolled to receive daratumumab and dexamethasone. Treatment cycles had a duration of 28 days. Subjects received treatment until either disease progression, death, unacceptable toxicity or for a maximum of 30 months. Drug administration and follow-up visits occurred more frequently for early cycles (weekly for the first 8 weeks, every two weeks for weeks 9-24 and then every 4 weeks). Disease evaluations occurred monthly and involved mainly measurements of myeloma proteins. Other assessments included bone marrow examinations, skeletal surveys, assessment of extramedullary plasmacytomas, and measurements of serum calcium corrected for albumin, and β2- microglobulin and albumin.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Voluntary written informed consent before performance of any study-related procedure.
3. Subject must have documented multiple myeloma as defined by the criteria below:

   Monoclonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma.

   AND any or more of the following myeloma defining events:
   * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

     * Hypercalcaemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL)
     * Renal insufficiency: creatinine clearance <40 mL per min or serum creatinine >177 μmol/L (>2 mg/dL)
     * Anaemia: haemoglobin value of >20 g/L below the lower limit of normal, or a haemoglobin value <100 g/L
     * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PETCT
   * Any one or more of the following biomarkers of malignancy:

     * Clonal bone marrow plasma cell percentage ≥60%
     * Involved:uninvolved serum free light chain ratio ≥100
     * >1 focal lesions on MRI studies
4. Prior treatment with at least two lines of treatment that included both bortezomib- and lenalidomide based regimens.
5. Documented evidence of progressive disease (PD) as defined by the modified IMWG criteria on or after the last regimen if the patient responded to previous regimens.
6. Subjects must have measurable disease as defined by any of the following:

   * Serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dL (except for IgA subtype: ≥ 0.5 g/dL) or urine M-protein level ≥ 200 mg/24 hours; or
   * Light chain multiple myeloma: Serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa lambda free-light-chain ratio.
7. Renal impairment defined as eGFR < 30 ml/min/1.73 m2 (calculated with the CKD-EPI formula) or in need for dialysis. Patients who undergo intraperitoneal dialysis may also be included.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.
9. Willingness and ability to participate in study procedures.
10. Reproductive Status

    1. Women of childbearing potential (WOCBP) must have two negative serum or urine pregnancy tests, one 10-14 days prior to start of the study drug and one within 24 hours prior to the start of study drug. Females are not of reproductive potential if they have been in natural menopause for at least 24 consecutive months, or have had a hysterectomy and/or bilateral oophorectomy.
    2. Women must not be breastfeeding.
    3. WOCBP must agree to follow instructions for methods of contraception for 4 weeks before the start of treatment with study drugs, for the duration of treatment with study drugs, and for 3 months after cessation of study treatment.
    4. Males who are sexually active must always use a latex or synthetic condom during any sexual contact with females of reproductive potential, even if they have undergone a successful vasectomy. They must also agree to follow instructions for methods of contraception for 4 weeks before the start of treatment with study drugs, for the duration of treatment with study drugs, and for a total of 3 months post-treatment completion.
    5. Male patients must not donate sperm for up to 90 days post treatment completion.
    6. Female patients must not donate eggs for up to 90 days post treatment completion.
    7. Azoospermic males and WOCBP who are not heterosexually active are exempt from contraceptive requirements. However, WOCBP will still undergo pregnancy testing as described in this section.

Exclusion Criteria:

1. Previous therapy with daratumumab or other anti-CD38 therapy.
2. Anti-myeloma treatment within 2 weeks prior to Cycle 1, Day 1.
3. Cumulative dose of corticosteroids greater than or equal to the equivalent of 140mg prednisone for ≥ 4 days or a dose of corticosteroids greater than or equal to the equivalent of 40 mg/day of dexamethasone for ≥ 4 days within the 2-week period prior to Cycle 1, Day 1.
4. Previous allogenic stem cell transplant; or Autologous Stem Cell Transplantation (ASCT) within 12 weeks before Cycle 1, Day 1.
5. Clinical signs of meningeal involvement of multiple myeloma.
6. Subject has either of the following:

   1. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
   2. Known moderate or severe persistent asthma (see Appendix 7), within 2 years from C1D1, or currently has uncontrolled asthma of any classification. Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
7. Clinically significant cardiac disease, including:

   1. Myocardial infarction within 1 year, or unstable or uncontrolled condition (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   2. Uncontrolled cardiac arrhythmia (CTCAE Grade 2 or higher) (atrial fibrillation with controlled ventricular rate is allowed) or clinically significant ECG abnormalities.
   3. ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
8. Any of the following:

   1. Known active hepatitis A
   2. Patient is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
   3. Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
9. Known to be seropositive for human immunodeficiency virus (HIV).
10. Amyloidosis, or any prior or concurrent malignancy, except for the following:

    1. Adequately treated basal cell or squamous cell skin cancer.
    2. Any cancer (other than in-situ) from which the subject has been disease-free for 3 years prior to study entry.
11. Any of the following laboratory test results during screening:

    1. Absolute neutrophil count ≤ 1.0 × 10^9/L;
    2. Hemoglobin level ≤ 7.5 g/dL (≤ 4.65 mmol/L);
    3. Platelet count < 75 × 10^9/L in patients in whom < 50% of bone marrow nucleated cells are plasma cells and < 50x10^9/L in patients in whom more than 50% of bone marrow nucleated cells are plasma cells;
    4. Alanine aminotransferase level ≥ 2.5 times the upper limit of normal (ULN);
12. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Kastritis, Assoc Prof, Principal Investigator — National and Kapodistrian University of Athens, School of Medicine, Athens, Greece
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Greece

REFERENCES:
- [Derived] Kastritis E, Terpos E, Symeonidis A, Labropoulou V, Delimpasi S, Mancuso K, Zamagni E, Katodritou E, Rivolti E, Kyrtsonis MC, Roussou M, Fotiou D, Theodorakakou F, Ntanasis-Stathopoulos I, Hatjiharissi E, Kanellias N, Migkou M, Cheliotis G, Manousou K, Gavriatopoulou M, Dimopoulos MA. Prospective phase 2 trial of daratumumab with dexamethasone in patients with relapsed/refractory multiple myeloma and severe renal impairment or on dialysis: The DARE study. Am J Hematol. 2023 Sep;98(9):E226-E229. doi: 10.1002/ajh.27001. Epub 2023 Jun 21. No abstract available. PMID 37340832

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD): Daratumumab:
  Daratumumab was given at a dose of 16 mg/kg administered as an intravenous (IV) infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Dexamethasone was administered according to the standard recommended dose of 40 mg (20 mg for patients > 75 years of age) orally once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle. Subjects received pre-infusion medications before infusions to mitigate potential infused-related reactions (IRRs).
  Dexamethasone:
  Dexamethasone was administered at 40 mg (20 mg for patients > 75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Started | 38
Completed | 15
Not Completed | 23
Not completed — Death | 17
Not completed — ICF withdrawal | 4
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD): Daratumumab:
  Daratumumab was given at a dose of 16 mg/kg administered as an intravenous (IV) infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Dexamethasone was administered according to the standard recommended dose of 40 mg (20 mg for patients>75 years of age) orally once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle. Subjects received pre-infusion medications before infusions to mitigate potential infused-related reactions (IRRs).
  Dexamethasone:
  Dexamethasone was administered at 40 mg (20 mg for patients >75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Greek | 32
  Other European | 4
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 34
  Italy | 4

OUTCOME MEASURES:

1. Primary Outcome: The Evaluation of Progression Free Survival (PFS) in Subjects With Relapsed or Refractory Multiple Myeloma and Renal Impairment Treated With Daratumumab and Dexamethasone.
Description: Progression free survival was defined as the time, in months, from treatment initiation (C1D1) to the date of the first documented disease progression or death due to any cause, whichever came first. Clinical deterioration was not considered progression. For patients who neither progressed nor died, the survival time was censored at the date of their last disease assessment. For patients who started a new anti-tumor treatment, survival time was censored at the date of the start of the new treatment.
Time Frame: Duration from first daratumumab administration until death or last assessment, months.
Population: Kaplan-Meier estimates for progression-free survival (PFS) in months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Months | 11.8 [2.8 to 20.8]
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; The PFS function was estimated using the Kaplan-Meier product-limit method. Median and two-sided confidence intervals (CIs) for PFS were computed and Kaplan-Meier plots of PFS were developed

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of subjects who achieve a best response of PR or better using modified IMWG criteria as their best overall response.
Time Frame: From first dose of Daratumumab until end of treatment, PD or death (approximately up to 30 months)
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Percent | 47.4 [31.5 to 63.2]
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Renal Response Rate (RRR)
Description: Renal response rate was defined as the proportion of enrolled subjects who achieve a best response of renal partial response (PRRenal) or better using the IMWG criteria.
Time Frame: From first dose of Daratumumab until end of treatment, PD or death (approximately up to 30 months )
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Percent | 18.4 [7.7 to 34.3]
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Duration of Response in Patients With RI
Description: Duration of response was restricted to the subjects that achieve a best objective response of PR or better. It was measured from the time, in months, that the criteria for objective response are first met until the date of a progression event (according to the primary definition of PFS).
Time Frame: Assessed monthly from first dose of Daratumumab until PD or death from any cause (approximately up to 30 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 18
Months | 28.4 [15.1 to NA] — The upper limit was not reached (NR).
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; The PFS function was estimated using the Kaplan-Meier product-limit method. Median and one-sided confidence intervals (CIs) for PFS were computed and Kaplan-Meier plots of PFS were developed

5. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy was defined as the time, in months, from Cycle 1 Day 1 to the date to next anti-neoplastic therapy or death from any cause, whichever comes first.
Time Frame: From first dose until the date to next anti-neoplastic therapy or death from any cause, whichever comes first (approximately up to 30 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Months | 18.0 [5.5 to NA] — The upper limit was never reached (NR).
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time, in months, from the first dose of therapy to the date of death from any cause.
Time Frame: Time from first dose of study treatment to death (approximately up to 30 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Months | 24.5 [5.5 to NA] — The upper limit was never reached (NR).
Statistical Analysis 1: Comparison: Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD); Test type: Other — The PFS function was estimated using the Kaplan-Meier product-limit method, a non-parametric statistic; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: To Assess the Safety and Tolerability of Daratumumab With Dexamethasone in Patients With Refractory and Relapsed Multiple Myeloma (RRMM) and Renal Impairment (RI).
Description: The incidence of Adverse Events and Treatment Emergent Adverse Events in patients with refractory and relapsed multiple myeloma and renal impairment treated with daratumumab with dexamethasone was assessed according to the common Terminology Criteria for Adverse Events.
Time Frame: Continuously throughout the study, starting from informed consent until 30 days after last study treatment (approximately up to 30 months).
Measure: Number; unit: Participants
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
Number analyzed (Participants) | 38
Participants
  Any (N)SAE | 34
  Any NSAE | 32
  Any SAE | 11
  Any (N)SADR related to daratumumab | 7
  Any NSADR related to daratumumab | 7
  Any SADR related to daratumumab | 1
  Any (N)SAE of Grade >=3 | 24
  Any (N)SAE of Grade 3 or 4 | 19
  Any fatal SAE | 7

ADVERSE EVENTS:
Time Frame: 3 years.
Description: The incidence of AEs was tabulated by the Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) and Preferred Term (PT), overall and by maximum Common Terminology Criteria for Adverse Events (CTCAE) grade.
Groups:
- Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD): Daratumumab:
  Daratumumab was given at a dose of 16 mg/kg administered as an intravenous (IV) infusion at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects received pre-infusion medications before infusions to mitigate potential infused-related reactions (IRRs).
  Dexamethasone:
  Dexamethasone was administered at 40 mg (20 mg for patients > 75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Arm/Group | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD)
All-Cause Mortality (participants affected / at risk) | 17/38
Serious Adverse Events (participants affected / at risk) | 11/38
Other Adverse Events (participants affected / at risk) | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD) (N=38)
Myocardial infarction (Cardiac disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 4
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial Receiving Daratumumab With Dexamethasone (DaraD) (N=38)
Anaemia (Blood and lymphatic system disorders) | 11
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 9
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 1
Swelling (General disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 5
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Tension (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03450057/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT03450057/SAP_001.pdf